CLINICAL TRIAL: NCT06735300
Title: Detection of Severe Acute Respiratory Syndrome Coronavirus 2 in Pregnant Women Treated with Nirmatrelvir/Ritonavir (Paxlovid) Using Saliva Polymerase Chain Reaction: a Prospective Cohort Study
Brief Title: Saliva PCR in Pregnant Women with COVID-19
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB: B-ER-111-164
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Coronavirus Disease 2019 (COVID-19) Pneumonia
Keywords: severe acute respiratory syndrome coronavirus 2; pregnancy; nirmatrelvir/ritonavir 25 (Paxlovid); saliva
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — nirmatrelvir; Ritonavir; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — nasopharyngeal specimens and saliva for RT-PCR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Nirmatrelvir/Ritonavir (Paxlovid) — After providing the potential benefits and associated risks of antiviral treatment with Paxlovid, patients made well-informed decisions about whether or not to receive Paxlovid (300/100 mg nirmatrelvir/ritonavir, Pfizer Inc., New York, NY, USA) twice daily for 5 days.

SUMMARY:
Abstract: Objectives We aim to study the relative viral load using saliva polymerase chain reaction among pregnant women treated with Paxlovid. Methods Pregnant women with coronavirus disease 2019 were allocated to two groups: those receiving Paxlovid and those receiving no antiviral agents. We compared the nasopharyngeal and salivary relative viral loads and their changes in saliva specimens. Results Among the 38 pregnant women, seventeen received Paxlovid, and 21 received no antiviral agents. The viral cycle threshold value of saliva was significantly higher than that from nasopharynx, with a median ± interquartile range of 26.44 ± 7.68 versus 17.6 ± 9.6 in the Paxlovid group (p = 0.005). Following treatment, the Paxlovid group showed a significant decrease in relative saliva viral load (cycle threshold value on Day 4/Day 5 minus Day 0) compared to the non-antiviral group (13.40 ± 5.64 versus -1.59 ± 9.63, p = 0.021). The detection rate of coronavirus disease 2019 using salivary polymerase chain reaction was 81.6% (31/38). Conclusions This study showed that saliva is a useful diagnostic tool for coronavirus disease 2019 in pregnant women, and a significant decrease in the relative viral load of saliva was observed in those treated with Paxlovid.

ELIGIBILITY:
Inclusion Criteria:

* This study enrolled pregnant women admitted to NCKUH 70 who tested positive for COVID-19 by real-time reverse transcription polymerase chain reaction (RT-PCR) of nasopharyngeal swab specimens. After providing the potential benefits and associated risks of antiviral treatment with Paxlovid, patients made a well-informed decision about whether or not to receive Paxlovid (300/100 mg nirmatrelvir/ritonavir, Pfizer Inc., USA) twice daily for 5 days.

Exclusion Criteria:

* Pregnant women were excluded if the time interval between the onset of symptoms and admission to our hospital was greater than seven days, in the case of insufficient saliva samples, or if any antiviral-related agents were administered, such as remdesivir, glucocorticoids, or interleukin-6 receptor antagonists.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From 1 June 2022 to 7 October 2022, 56 pregnant women were screened for eligibility, of which 38 were included in the analysis. Of these, 17 pregnant women were administered Paxlovid, and 21 pregnant women were not administered any antiviral treatment. The two groups of pregnant women were comparable across the two cohorts, except for an earlier gestational age at diagnosis of COVID-19 in the Paxlovid group than in the non-antiviral group (35.4 weeks versus 37.5 weeks, p = 0.022). Among women treated with Paxlovid, 47.1% had gestational complications compared with 9.5% of those without antiviral treatment (p = 0.012).
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Salivary viral load | From enrollment to the end of treatment at 7 days
  The amount of decrease in salivary viral load after taking Paxlovid

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng 68 Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No